CLINICAL TRIAL: NCT02071329
Title: A Randomised, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Efficacy and Immunogenicity of an Influenza A Vaccine (Vaccine FP-01.1) in Healthy Volunteers Following Virus Challenge
Brief Title: Safety, Tolerability, Efficacy and Immunogenicity of an Influenza A Vaccine (FP-01.1) in Healthy Volunteers Following Virus Challenge
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immune Targeting Systems Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FP-01.1_CS_04; 2013-004612-22 (EudraCT Number)
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Influenza A
Keywords: FP-01.1; Influenza A; Flu; Vaccine; Virus; H1N1; Challenge
MeSH Terms: conditions — Influenza, Human; Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaccine FP-01.1 (Experimental): Vaccine FP-01.1
  Interventions: Drug: Vaccine FP-01.1; Other: Virus Challenge
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo; Other: Virus Challenge

INTERVENTIONS:
Drug: Vaccine FP-01.1
  Arms: Vaccine FP-01.1
Drug: Placebo
  Arms: Placebo
Other: Virus Challenge
  Other Names: Live, wild-type A/California/H1N1 2009

SUMMARY:
The purpose of this study is to assess the safety, tolerability, efficacy, and immunogenicity of an influenza A vaccine (vaccine: FP-01.1), as compared to placebo, in healthy volunteers following a dose of influenza A virus.

DETAILED DESCRIPTION:
This study is designed to further investigate the safety and tolerability of FP-01.1 in healthy subjects and to explore the effect of prior vaccination with Vaccine FP-01.1 (250 μg/peptide) or placebo on the incidence, severity and duration of the signs and symptoms of influenza and the magnitude of viral load in nasal secretions and duration of viral shedding, after challenge with an A/California/H1N1 2009 influenza virus, in healthy male and female subjects. The study will also be used to provide additional information on the immunological responses (both humoral and cell-mediated immune [CMI] responses) following Vaccine FP-01.1 treatment and to investigate potential markers for protection against influenza A infection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 45 years inclusive, with a body mass index of 18.0 to 32.0 kg/m2 inclusive and body weight of 50.0 to 110.0 kg inclusive;
2. Subjects who are able and willing to give written informed consent to participate;
3. Healthy, as determined by medical history, physical examination, vital signs, 12-lead ECG, and clinical safety laboratory examinations at screening (Visit 2) and Day C-1 (prior to virus challenge), as determined by the Investigator;
4. Absent or low levels of detectable pre-existing antibodies to the challenge H1N1 virus (HI titre of ≤10) and predicted seasonal H3N2 virus (HI titre of ≤40) prior to vaccination;
5. Subjects who are non-smokers for at least 3 months preceding screening (Visit 2) and able to refrain from smoking until after the completion of Visit 9 [Day C29]);
6. Females of non-childbearing potential or female subjects of childbearing potential who are using 2 medically acceptable methods of contraception;
7. Comprehension of the study requirements, expressed availability for the required study period, and ability to be quarantined for up to 10 days and to attend the scheduled follow-up visits (Day C29 and Day 209);
8. Negative alcohol and urine drug screening tests on screening and prior to entering quarantine (Day C-1);
9. Being willing to adhere to the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

1. Subjects who do not conform to the above inclusion criteria;
2. Receipt of any influenza vaccine after 31 August 2011;
3. Significant adulthood history of seasonal hay fever or a seasonal allergic rhinitis or perennial allergic rhinitis or chronic or nasal or sinus condition such as chronic sinusitis;
4. Abnormal nasal structure including septal deviation and nasal polyps;
5. History of asthma (childhood asthma allowed), bronchiectasis, emphysema, chronic obstructive pulmonary disease or any other chronic lung disease in the last 10 years;
6. Current use or use within the last 7 days from screening day (Visit 2) of intranasal corticosteroids;
7. Subjects who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiac/cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders; this includes, but is not limited to, institution of new surgical or medical treatment (for a chronic condition), or a significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months of screening and reconfirmed before first vaccination;
8. Subjects who do not agree to use medically acceptable methods of contraception;
9. Female subjects who are pregnant, trying to become pregnant or are breast feeding;
10. Diastolic blood pressure <50 or >90 mmHg, a systolic blood pressure <100 or >150 mmHg, a pulse <40 or >100 beats per minute (bpm) after resting for 5 minutes;
11. Forced expiratory volume at one second (FEV1) ≤90% of predicted FEV1;
12. Blood haemoglobin A1c >6.0%;
13. Positive serology for human immunodeficiency virus (HIV) 1 or HIV 2, hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies;
14. Cancer or treatment for cancer, within 5 years of Visit 2, excluding basal cell carcinoma of the skin, which is allowed;
15. Presence of immunosuppression or any medical condition that may be associated with impaired immune responsiveness, including, but not limited to, diabetes mellitus and inflammatory bowel disease;
16. Presently receiving or a history of receiving during the 3-month period prior to screening, any medications or other treatments that may adversely affect the immune system such as allergy injections, immune globulin, interferon (IFN), immunomodulators, cytotoxic drugs or other drugs known to be frequently associated with significant major organ toxicity, or systemic corticosteroids (oral or injectable) azathioprine or mercaptopurine; topical corticosteroids, except intranasal, will be allowed;
17. Anticipated presence of a household contact with documented severe immunosuppression (including but not limited to HIV, anyone who has haematological malignancy or is taking immunosuppressant medication), either as a result of disease and/or therapy within 2 weeks following discharge from the virus challenge quarantine period;
18. Anticipated presence of a household contact age 5 years or younger, within 2 weeks following discharge from the virus challenge quarantine period;
19. Anticipated presence of a household contact age 65 years or older, within 2 weeks following discharge from the virus challenge quarantine period;
20. Anticipated presence of a household contact with diagnosed emphysema, chronic obstructive pulmonary disease, severe lung disease or any organ or bone marrow transplant, within 2 weeks following discharge from the virus challenge quarantine period;
21. Current professional activity as a carer or healthcare worker;
22. Anticipated presence of a pregnant household contact, within 2 weeks following discharge from the virus challenge quarantine period;
23. History of Guillain-Barré syndrome;
24. History of drug or chemical/alcohol abuse in the year before the study (Visit 2);
25. Receipt of any investigational virus product or any investigational product (IMP) within 3 months prior to first vaccination, or currently enrolled in any investigational drug study or intends to enrol in such a study within the ensuing study period;
26. Receipt of blood or blood products 6 months prior to first vaccination or planned administration during the study period;
27. Blood donation in the 3 months prior to screening (Visit 2);
28. Acute disease within 72 hours prior to vaccination, defined as the presence of a moderate or severe illness with or without fever (as determined by the Investigator through medical history and physical examination), or presence of a fever (>37.7ºC oral temperature);
29. Elevated white cell count >9.5 x 109/L, absolute neutrophil count >6.9 x 109/L or serum C-reactive protein concentration >10.0 mg/L at screening (Visit 2) or Day C-1;
30. Any condition that, in the opinion of the Investigator, might interfere with the primary study objective;
31. Known or suspected intolerance or hypersensitivity to the IMP or closely related compounds, known allergy to egg or egg protein or any of the stated excipients;
32. Known or suspected intolerance or hypersensitivity to Tamiflu or Relenza;
33. Subject with suspected recent (≤6 months) experience of influenza-like illness (fever [>37.7ºC] and cough and/or sore throat >2 days, in the absence of a known cause other than influenza);
34. Subjects who have significant scarring, tattoos, abrasions, cuts or infections, that in the opinion of the Investigator could interfere with evaluation of injection site local reactions, over the deltoid region of both arms as these will be the dose site;
35. Subjects who are vegans or have medical dietary restrictions;
36. Subjects who cannot communicate reliably with the Investigator.

Exclusion Criteria for Virus Challenge

Randomised subjects who have completed the vaccination phase of the study (Day 1 to Day 36) will be excluded from proceeding to the virus challenge part of the study under the following conditions:

* Subjects have not received 2 administrations of Vaccine FP-01.1 or placebo per protocol;
* Positive HI titre on Day 29 (defined as HI titre >20 for the H1N1 challenge virus);
* Presence of any mild, moderate or severe influenza symptoms or signs as assessed by the subject scoring card or targeted physical examination prior to dosing;
* An oral temperature >37.7°C on Day C-1 or Day C1 prior to dosing.

Any subjects who meet the criteria listed above must not be challenged.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety | Day 1 - 72
  The safety evaluation will include adverse events (AEs), clinical laboratory safety tests, physical examinations, vital signs, 12-lead ECG parameters, spirometry and local injection site reactions.

SECONDARY OUTCOMES:
Efficacy | Day 44 - 52
  To compare the incidence, severity and duration of signs and symptoms of influenza-like illness after virus challenge between subjects pre-vaccinated with Vaccine FP-01.1 and subjects pre-vaccinated with placebo.
Pharmacodynamics | Day 45 -52
  To compare the incidence, magnitude and duration of viral shedding after virus challenge between subjects pre-vaccinated with Vaccine FP-01.1 and subjects pre-vaccinated with placebo.
Immunogenicity | Day 1-72
  To assess magnitude, breadth and kinetics of immune response to FP-01.1

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles Drug Research Unit at Guy's Hospital, London, United Kingdom